CLINICAL TRIAL: NCT06389110
Title: Phase III Clinical Study to Evaluate the Efficacy of Alleance® (Atropine Sulfate 0.01%) as a Treatment to Delay the Progression of Myopia and Axial Ocular Elongation in Children.
Brief Title: Study to Evaluate the Efficacy of Alleance® (Atropine Sulfate 0.01%) as a Treatment to Delay Myopia and Axial Ocular Elongation in Children.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOPH201-1023/III
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Myopia; Myopia, Progressive
MeSH Terms: conditions — Myopia; Myopia, Degenerative

STUDY DESIGN:
Intervention Model Description: This is a study to demonstrate superiority, double-blind, randomized, controlled, comparative, and multicenter phase III clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alleance® (Active Comparator): Alleance®. Atropine sulfate 0.01%. Ophthalmic solution.
  * Dosage: 1 drop QD [1] (once a day), at night, for 12 months.
  * Route of administration: Ophthalmic
  Interventions: Drug: Alleance®
- Placebo (Placebo Comparator): * Placebo. Ophthalmic solution.
  * Dosage: 1 drop QD [1] (once a day), at night, for 12 months.
  * Route of administration: Ophthalmic
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alleance® — Atropine sulfate 0.01%, ophthalmic solution.
  Arms: Alleance®
Drug: Placebo — Ophthalmic solution.
  Arms: Placebo

SUMMARY:
Phase III clinical study to evaluate the efficacy of Alleance® (atropine sulfate 0.01%) ophthalmic solution through the incidence of unexpected adverse events, changes in Best Corrected Visual Acuity (BCVA), changes in intraocular pressure, changes in the amplitude of accommodation, compared to placebo, as a treatment to delay the progression of myopia and axial ocular elongation in children.

DETAILED DESCRIPTION:
This is a study to demonstrate superiority, double-blind, randomized, controlled, comparative, and multicenter phase III clinical trial.

Primary Objective:

- To demonstrate the superiority of Alleance® compared to placebo in delaying myopia progression in children.

Specific objectives:

* To demonstrate the reduction in progression in spherical equivalent in children using Alleance® compared to placebo after 12 months of treatment.
* To demonstrate the reduction in progression in ocular axial length in children using Alleance® compared to placebo, after 12 months of treatment.

Secondary objectives:

* To compare the incidence of adverse events related to the interventions.
* Compare the incidence of photophobia between interventions.
* To assess pupillary diameter between the interventions.
* To assess best-corrected far visual acuity between interventions.
* To assess near best-corrected visual acuity between interventions.
* To assess the amplitude of accommodation between interventions.
* Assess intraocular pressure (IOP) between procedures.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 3 to 12 years
* Male or female sex.
* The parent(s) or legal guardian(s) must voluntarily give their signed informed consent.
* From the age of 7 years and older, the subject's willingness to participate in the research study will be expressed in writing. In the case of subjects under 7 years of age, only the signature of the informed consent by the parent(s) or legal guardian(s) will be required, provided that the subject's verbally expressed will is respected.
* Ability and willingness to comply with the scheduled visits, treatment plan and other study procedures.
* Female subjects, who have already presented their menarche, must have a negative urine pregnancy test at the time of screening.
* Female subjects who have already experienced menarche should secure a method of contraception for the duration of the study. Acceptable contraceptive methods include abstinence (defined as abstinence from heterosexual intercourse from study entry until completion) or use of a highly effective contraceptive method, including hormonal contraception, barrier methods or intrauterine device).
* Refractive error of spherical equivalent between -0.50 to -6.00 D in each eye, measured by autorefraction and cycloplegic retinoscopy.
* Astigmatism less than -1.50 D in each eye, measured by autorefraction and retinoscopy.
* Spherical equivalent anisometropia ≤ 1.50 D measured by autorefraction and cycloplegic retinoscopy.
* Best corrected visual acuity (BCVA) normal for age.
* Normal binocular function and stereopsis for age.
* Normal intraocular pressure (< 21 mmHg).
* Gestational age ≥ 32 weeks and birth weight > 1500 g.

Exclusion Criteria:

* Allergy to atropine or any of the components of the investigational products.
* Previous or current use of atropine, orthokeratology lens or other optical methods for myopia control (bifocal, progressive, multifocal, or defocusing air or contact lenses). Only prior or current use of frame lenses or monofocal contact lenses for the correction of myopic or myopic/astigmatic refractive error will be allowed.

History or current history of amblyopia or manifest strabismus, including intermittent tropia.

* Heart rate > 120 beats per minute persistently (for more than 10 minutes) at the time of screening/baseline visit.
* History of any disease or syndrome predisposing the subject to severe myopia (Marfan syndrome, Stickler syndrome, retinopathy of prematurity, etc.).
* History of serious systemic disease that, in the investigator's judgment, would make the subject ineligible (e.g., cardiac, endocrine, respiratory, neurologic [infantile cerebral palsy], Down syndrome, etc.).
* History or current history of glaucoma or ocular hypertension.
* History of any refractive ocular anatomical anomaly (keratoconus, lenticonus, spherophakia, aphakia, etc.).
* History of ocular diseases, excluding myopia (corneal alterations/opacities, cataract, retinal alterations, inflammatory diseases, etc.).
* History of any type of ocular surgery.
* For female subjects who have presented their menarche: being pregnant or breastfeeding.
* Having participated in clinical research studies 30 days prior to inclusion in the present study.
* Previous participation in this study.
* Present unresolved ocular lesions or trauma at the time of study entry.
* Present active inflammatory or infectious ocular disease at the time of study entry.
* Having undergone surgical procedures, not ophthalmologic, within the last 3 months.
* Chronic use of any topical or systemic antimuscarinic/anticholinergic medication (atropine, scopolamine, tropicamide) within 21 days prior to screening, and/or anticipated need for its chronic use during the study period (more than 7 consecutive days in a month or more than 30 days total in a year). The use of cycloplegic drops for ophthalmologic examination is allowed.
* Be or have an immediate family member (e.g., parent/legal guardian or sibling) who is part of the research site or sponsor´s staff.

Elimination Criteria:

* Withdrawal of their consent to participate in the study (informed consent form).
* Occurrence of a serious adverse event, whether related or not to the interventions, that in the opinion of the principal investigator (PI) and/or the sponsor, could affect the patient's fitness to safely continue with the study procedures.
* Non-tolerability or hypersensitivity to any of the compounds used during the tests -(fluorescein, tetracaine).
* Non-tolerability or hypersensitivity to any of the drugs under investigation.
* Adherence < 80% determined by the subject's diary and corroborated by the final weight of the research products (RP) compared to the initial weight.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 123 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the spherical equivalent | Days 0 (Basal visit), 14 (Visit 1), 45 (Safety call 1), 180 (Visit 3), 225 (Safety call 2), 270(Visit 4), 315 (Safety call 4), 365 (Final Visit), 380 (Last Final Safety call)
  The reduction in progression in spherical equivalent, will be calculated by combining the spherical component (E) and the cylindrical component (C) of the refractive error, independently for each eye: EE=E+C2
Changes in axial eye length | Days 0 (Basal visit), 14 (Visit 1), 45 (Safety call 1), 180 (Visit 3), 225 (Safety call 2), 270(Visit 4), 315 (Safety call 4), 365 (Final Visit), 380 (Last Final Safety call)
  The reduction in progression in ocular axial length will be measured utilizing optical biometry.

SECONDARY OUTCOMES:
Incidence of unexpected adverse events related to the interventions | Days 0 (Basal visit), 14 (Visit 1), 45 (Safety call 1), 180 (Visit 3), 225 (Safety call 2), 270(Visit 4), 315 (Safety call 4), 365 (Final Visit), 380 (Last Final Safety call)
  Any unfavorable medical condition affecting the subject after the administration of the investigation product, related to such intervention.
Incidence of photophobia between interventions | Days 0 (Basal visit), 14 (Visit 1), 180 (Visit 3), 365 (Final Visit), 380 (Last Final Safety call)
  Any signs of uncomfortable vision, based on the diffusion of light through the ocular media or on a transient or permanent lack of adaptation. The subjects will be questioned regarding this symptoms' incidence.
Changes in pupillary diameter between the interventions | Days 0 (Basal visit), 14 (Visit 1), 180 (Visit 3), 365 (Final Visit), 380 (Last Final Safety call)
  The changes in pupillary diameter will be evaluated through the optical biometer or by the OPD scan Topographer III®.
Changes in Best Corrected Visual Acuity (BCVA) | Days 0 (Basal visit), 14 (Visit 1), 180 (Visit 3), 365 (Final Visit), 380 (Last Final Safety call)
  The best corrected visual acuity will be evaluated through the Snellen chart in subjects ≥ 6 years of age.
  The LEA chart is used to assess visual acuity in children older than 30 months of age.
Changes in near best-corrected visual acuity | Days 0 (Basal visit), 14 (Visit 1), 180 (Visit 3), 365 (Final Visit), 380 (Last Final Safety call)
  The bear best corrected visual acuity will be evaluated through the LEA chart, in subjects ≤ 5 years of age. The bear best corrected visual acuity will be evaluated through the Snellen chart in subjects ≥ 6 years of age.
  The LEA chart is used to assess visual acuity in children older than 30 months of age
Changes in the amplitude of accommodation (AA) between interventions | Days 0 (Basal visit), 14 (Visit 1), 180 (Visit 3), 365 (Final Visit), 380 (Last Final Safety call)
  The amplitude of accommodation(AA) is the difference between the resting state of the crystalline lens (far point) and the maximum refractive focus in diopters that the emmetropic or emmetropic patient can use to focus on near objects.
  The AA will be measured by the Donders method or by the approach method, utilizing the LEA chart.
Changes in intraocular pressure (IOP) | Days 0 (Basal visit), 14 (Visit 1), 180 (Visit 3), 365 (Final Visit), 380 (Last Final Safety call)
  Previous instillation of topical anesthetic, the IOP (both eyes) will be measured through a Goldmann tonometer during visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Innovación Y Desarrollo En Ciencias de La Salud S de Rl de Cv, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No